CLINICAL TRIAL: NCT03419377
Title: Lichen Sclerosus - the Influence on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Research Coordinator, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHN_DMK_02
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Lichen Sclerosus
Keywords: Treatment; Quality of Life; Sexology; Women
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care and sexological counseling (Experimental): Standard care including gynecological examination and 6-8 sexological consultations.
  Interventions: Other: Standard care and sexological counseling
- Standard care (No Intervention): Standard care including gynecological examination.

INTERVENTIONS:
Other: Standard care and sexological counseling — 6-8 sexological consultants in a period of six months
  Arms: Standard care and sexological counseling

SUMMARY:
A randomised controlled trial of Lichen Sclerosus in a period of six months measuring Quality of Life and sexuality among women with Lichen Sclerosus.

DETAILED DESCRIPTION:
The patients are randomized to an intervention Group and a control Group. The intervention gets 6-8 visits with clinical sexologist and the control Group is having the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Lichen Sclerosus
* Age over 18 years

Exclusion Criteria:

* Patients who does not understand or speak Danish
* Patients with a psychiatric diagnosis and can not follow the course

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Quality of Life in women with Lichen Sclerosus | Six months
  Change in EuroQol five dimension (EQ-5D) score. The descriptive system comprises 5 dimensions (mobili-ty, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The answers given to EQ-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.

CONTACTS AND LOCATIONS:
Locations (1):
- Vendsyssel Hospital, Hjørring, Denmark

REFERENCES:
- [Derived] Vittrup G, Westmark S, Riis J, Morup L, Heilesen T, Jensen D, Melgaard D. The Impact of Psychosexual Counseling in Women With Lichen Sclerosus: A Randomized Controlled Trial. J Low Genit Tract Dis. 2022 Jul 1;26(3):258-264. doi: 10.1097/LGT.0000000000000669. Epub 2022 Mar 25. PMID 35333024